CLINICAL TRIAL: NCT00981669
Title: Evaluation of Rotavirus Vaccine Produced by Butantan Institute. Phase I - Safety, Tolerability and Immunogenicity Evaluation
Brief Title: Rotavirus Vaccine Produced by Butantan Institute
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1242/06
Record Dates: First submitted 2009-09-17; First posted 2009-09-22 (Estimated); Results first posted 2013-04-25 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-03

CONDITIONS: Rotavirus Infections
Keywords: brazilian pentavalent rotavirus vaccine; safety; tolerability; immunogenicity
MeSH Terms: conditions — Rotavirus Infections | interventions — Rotavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rotavirus vaccine (Experimental): 3 doses with 6 weeks interval
  Interventions: Biological: rotavirus vaccine
- placebo (Placebo Comparator): 3 doses with 6 weeks interval
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: rotavirus vaccine — 3 doses with 6 weeks interval
  Other Names: brazilian rotavirus vaccine
  Arms: rotavirus vaccine
Biological: placebo — 3 doses with 6 weeks interval
  Other Names: butantan placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to describe the safety, tolerability and immunogenicity of the pentavalent rotavirus vaccine produced by Butantan Institute.

DETAILED DESCRIPTION:
The Brazilian National Immunization Program (PNI) has introduced a oral monovalent vaccine against rotavirus for infants in its immunization schedule since 2006. Its introduction increased the Brazilian Ministry of Health budget because the vaccination in Brazil is free of charge. An agreement between Path Foundation and Butantan Institute has made possible the transfer of technology to Butantan Institute to produce, at a reduced cost, a pentavalent rotavirus vaccine including the the rotavirus serotypes more frequent in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Male healthy
* Age ≥18-40 years
* Not taking immunosuppressive drugs
* No clinical history of gastrointestinal diseases or surgeries
* No history of cardiac, neurologic, immunologic or endocrine diseases
* Normal eligibility laboratory tests
* To be willing to participate and sign the informed consent form
* No participation in another clinical trial in the past 6 months

Exclusion Criteria:

* Had received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander R Precioso, MD,PhD, Study Director — Butantan Institute
Locations (1):
- Instituto da Criança do Hospital das Clinicas da Faculade de Medicina da USP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Higashi HG, Luna E, Precioso AR, Vilela M, Kubrusly FS, Dias WO, Raw I. Acellular and "low" pertussis vaccines: adverse events and the role of mutations. Rev Inst Med Trop Sao Paulo. 2009 May-Jun;51(3):131-4. doi: 10.1590/s0036-46652009000300002. PMID 19551286

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: From February to August 2009.79 healthy adult volunteers from 18 to 40 years of age were selected. Participants were screened for eligibility and enrolled by the investigators following the signing of an informed consent. Due to a recommendation from ANVISA, female volunteers were not allowed to be recruited.
Pre-assignment Details: 98 potential volunteers were interviewed, 80 of them were enrolled: 40 volunteers were allocated to receive the investigational product (rotavirus vaccine) and 40 were allocated to receive placebo; 79 completed the follow-up. Before randomization 18 volunteers were excluded, 3 refused to participate and 15 had screening failure
Period: Overall Study
Arm/Group | Rotavirus Vaccine | Placebo
Started | 40 | 40
Completed | 39 | 40
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: In the vaccine gorup one volunteer was not considered for the final analysis because He received the second dose of the vaccine in an anapropriate interval.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotavirus Vaccine | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.2 (6.6) | 28.2 (6.2) | 28.7 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 40 | 40 | 80
Region of Enrollment [Number; unit: participants]
  Brazil | 40 | 40 | 80

OUTCOME MEASURES:

1. Secondary Outcome: Anti-rotavirus IgA Level.
Description: It was evaluated by anti-rotavirus IgA levels in terms of optical density. Pre-vaccination levels of anti-rotavirus antibodies were not considered as an exclusion criterion. Seroconversion was considered as a fourfold increase in IgA titers. The proportion of seroconverters in both groups was compared. IgA levels in optical density were not converted to any unit of measure.
Time Frame: before each dose (total of doses:3) and after 6 weeks of the third dose
Population: As in most phase I trials, sample size was not calculated to provide statistically significant differences between groups. Rather, a descriptive analysis on the frequency of AE and immunogenicity data was undertaken.
Measure: Median (Inter-Quartile Range); unit: Arbitrary units
Arm/Group | Rotavirus Vaccine | Placebo
Number analyzed (Participants) | 39 | 40
Arbitrary units | 0.51 [0.41 to 0.71] | 0.35 [0.30 to 0.46]

2. Primary Outcome: Number of Participants With Adverse Events.
Description: Safety and tolerability were evaluated by monitoring occurence of fever, diarrhea, vomiting, abdominal pain and increase of liver enzymes.
Time Frame: Within the first five days post-vaccination.
Measure: Number; unit: participants
Arm/Group | Rotavirus Vaccine | Placebo
Number analyzed (Participants) | 39 | 40
participants | 14 | 12

ADVERSE EVENTS:
Time Frame: Complaints and solicited symptoms were investigated following the first five days after vaccination.
Arm/Group | Rotavirus Vaccine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 10/39 | 9/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotavirus Vaccine (N=39) | Placebo (N=40)
Headache (Nervous system disorders) | 3 (3) | 2 (2)
Gastrointestinal Symptoms (Gastrointestinal disorders) | 5 (5) | 7 (7)
Loss of appetite (General disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The vaccine candidate needs to be evaluated further in larger trials, among the target population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes